CLINICAL TRIAL: NCT05634551
Title: Perceptions on Expected Outcomes of Immunotherapy in Advanced Cancer Patients With Poor Performance Status
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Conquer Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0348; NCI-2022-09969 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Questionnaires (All Participants): If participants are found to be eligible and agree to take part in the study, information about you (such as age, gender, race, ethnicity, marital status, education, employment status, religious beliefs, and information about your cancer diagnosis and history, current therapy and goal of cancer therapy) will be collected.
  Interventions: Behavioral: Questionnaires
- Interview (Some Participants): Not every participant will be asked to have an interview. It is expected that about 20-30 participants will take part in the interview part of the study.
  Interventions: Behavioral: Interview

INTERVENTIONS:
Behavioral: Questionnaires — Participants will complete 5 questionnaires about any symptoms participants may be having, any anxiety and/or depression participants may be having, your preference in decision-making, and your expectations about your treatment. It should take about 30 minutes to complete all 5 questionnaires
  Groups: Questionnaires (All Participants)
Behavioral: Interview — The interview will last about 30-45 minutes. The interview will be conducted over the phone or remotely over Zoom or FaceTime (based on your preference)
  Groups: Interview (Some Participants)

SUMMARY:
To better understand your feelings and expectations about immunotherapy

DETAILED DESCRIPTION:
Primary Objective:

1. To compare expectations of survival benefit from immunotherapy between advanced cancer patients with poor performance status (PS) and their oncologists. We hypothesize that, compared to their oncologists, patients will have expectations for greater likelihood of survival beyond 2 years.

Secondary Objectives:

1. To compare expectations of therapeutic benefit of immunotherapy between advanced cancer patients with poor PS and their oncologists. We hypothesize that, compared to their oncologists, patients will have expectations for greater likelihood of cure, quality of life improvement, and lower likelihood of adverse events.
2. To qualitatively describe the priorities and preferences for information of advanced cancer patients with poor PS when considering immunotherapy treatment.
3. To evaluate the associations between discrepant expectations with patients' sociodemographic and clinical characteristics.
4. To compare patient and oncologist expectations with actual treatment outcomes and survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patients being considered for or within 2 months of starting immunotherapy for advanced cancer
2. Patient ≥18 years of age
3. ECOG ≥2
4. Cognitively able to understand consent and complete questionnaire as determined by the interviewer at the time of study enrollment
5. English speaking
6. Willing to participate in the study and sign informed consent
7. The study will include medical oncologists that treat advanced cancers

Exclusion Criteria:

1. Treatment for curative intent
2. Presence of Delirium (as determined by score >13 on MDAS 46, appendix A)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: M D Anderson Cancer
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-08-02 (Actual)

PRIMARY OUTCOMES:
Discrepancy in expectation of survival for 2 years or more between the patient and oncologist | through study completion; an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Yennu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org